CLINICAL TRIAL: NCT00507975
Title: Assessment of the Effectiveness of Nicotine Replacement Therapies (Nicotine Patches Delivering Nicotine 16 h/24 h) in 400 Pregnant Smokers. Randomized, Placebo-controlled, Multicenter, National Study. The SNIPP.
Brief Title: Study of Nicotine Patch in Pregnancy (SNIPP)
Acronym: SNIPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P060604
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2007-07

CONDITIONS: Smoking
Keywords: Smoking; pregnancy; newborn; birth weight; nicotine patch; birth
MeSH Terms: conditions — Smoking; Birth Weight

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): The main aim of this study is to assess the effectiveness of nicotine patch comparatively to a placebo patch in pregnant women on birth weight and maternal smoking abstinence. The main secondary objective is the assessment of safety of these treatments for the fetus/newborn and for the mother.
  Interventions: Drug: nicotine versus placebo
- B (Experimental): The main aim of this study is to assess the effectiveness of nicotine patch comparatively to a placebo patch in pregnant women on birth weight and maternal smoking abstinence. The main secondary objective is the assessment of safety of these treatments for the fetus/newborn and for the mother.
  Interventions: Drug: nicotine versus placebo

INTERVENTIONS:
Drug: nicotine versus placebo — The main aim of this study is to assess the effectiveness of nicotine patch comparatively to a placebo patch in pregnant women on birth weight and maternal smoking abstinence. The main secondary objective is the assessment of safety of these treatments for the fetus/newborn and for the mother.

SUMMARY:
There are no established evidences as to the effectiveness in smoking pregnant women of nicotine patches in increasing birth weight, smoking abstinence during pregnancy and concerning the safety their for the fetus/newborn. Moreover, recent studies have shown that the metabolism of nicotine is speeded up in pregnant women suggesting that dose adaptation may be necessary in this population. The main aim of this study is to assess the effectiveness of nicotine patch comparatively to a placebo patch in pregnant women on birth weight and maternal smoking abstinence. The main secondary objective is the assessment of safety of these treatments for the fetus/newborn and for the mother.

DETAILED DESCRIPTION:
Smoking during pregnancy is one of the main causes of low birth weight and several disorders during pregnancy involving the mother, the fetus/newborn or both. Only one previous study assessed the efficacy of 16 hours nicotine patch proposed for 3 months in pregnant women for smoking cessation. This study seemed to be underpowered and the compliance was very poor. However, some benefit on birth weight was observed.

The aim of the present study is to demonstrate whether nicotine replacement therapy with 16 h nicotine patch every day increases or not birth weight and abstinence during pregnancy in smoking women. Secondarily, it is aimed to provide descriptive information about the safety of nicotine patches in pregnant women.

This is a double blind, randomized, placebo controlled study. With 200 pregnant women in each arm it will have sufficient power to conclude about differences in birth weight and maternal abstinence between nicotine and placebo.

Women are recruited by health care professionals and directed to the obstetrical departments having previously been agreed to participate in the study.

After a grace period of one month without pharmacological treatment, the pregnant women are randomized into the placebo (N=200) or the nicotine group (N=200). Treatment duration is from randomization till delivery meaning a maximum length of drug/placebo exposure of 6 month during pregnancy. No treatment is started earlier than 3 months' pregnancy. Women may optionally continue their treatment for at least up to 2 months after birth.

At the inclusion visit when the women are smoking, saliva cotinine is collected and determined. The first dose of nicotine is adapted according to the saliva cotinine when smoking to obtain approximately 100 % substitution. A second saliva cotinine determination is realized 2 weeks later and at the next visit nicotine's daily dose is determined according to this second saliva cotinine results for the whole duration of pregnancy. This dose-adaptation is necessary to avoid as far as possible under- and overdosing of nicotine.

The women undergo monthly visits as it is usual and recommended in France. They are followed as well as their newborn up to 2 months after birth.

During the visits standard obstetrical information along with smoking related information and the routinely realized echography data are recorded and birth characteristics collected.

In a subgroup of pregnant women having given their written informed consent and undergoing an amniocentesis for medical reasons, nicotine and cotinine in amniotic fluid will be determined.

In a subgroup of pregnant women having given their written informed consent and breast feeding their baby during the 2 months period after birth, nicotine and cotinine in maternal milk are determined.

There are 2 main outcome comparisons between the nicotine patch and the placebo patch groups: birth weight and maternal continuous, complete abstinence during pregnancy

ELIGIBILITY:
Inclusion Criteria:

* smoking pregnant woman unable to quit smoking during the first 3 months of pregnancy
* smoking ≥ 5 cigaret/day despite standard medical advice and cognitive-behavioral counselling
* aged ≥ 18 years
* health insured
* motivated to stop smoking; motivation score ≥ 5 on a scale ranging from 0 to 10
* amenorrhea of 9 to 20 weeks
* having signed the written informed consent

Exclusion Criteria:

* non-pregnant women
* men

Pregnant woman:

* who does not agree to use a nicotine or placebo patch
* with presence of chronic psychiatric comorbidity treated continuously by antidepressant, neuroleptic or anxiolytic
* with skin disorder contraindicating the use of a transdermal patch
* with known hypersensitivity to transdermal patch or to one of its constituents
* using other nicotine containing pharmaceutical products (gum, lozenge, inhaler, sublingual tablets)
* using other forms of tobacco than cigaret (cigaret, pipe or any form of smokeless tobacco)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 404 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Continuous and complete smoking abstinence of the pregnant women from the first administration of nicotine/placebo patch until delivery. | from the first administration of nicotine/placebo patch until delivery

SECONDARY OUTCOMES:
All adverse events occurring during pregnancy | during pregnancy
Point prevalence (7-days) smoking abstinence | 7-days smoking abstinence
Vital signs of the mother and her body weight | during pregnancy
Echography results of the foetus | during the pregnancy
Birth characteristics of the newborn (Apgar, head circumference, height) | at the delivery
Compliance with treatment | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Ivan BERLIN, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Groupe Hospitalier Pitié-Salpétrière, Unité de Recherche Clinique, Paris
  - Hopital La Pitie Salpetriere, Paris

REFERENCES:
- [Result] Wisborg K, Henriksen TB, Jespersen LB, Secher NJ. Nicotine patches for pregnant smokers: a randomized controlled study. Obstet Gynecol. 2000 Dec;96(6):967-71. doi: 10.1016/s0029-7844(00)01071-1. PMID 11084187
- [Result] Benowitz N, Dempsey D. Pharmacotherapy for smoking cessation during pregnancy. Nicotine Tob Res. 2004 Apr;6 Suppl 2:S189-202. doi: 10.1080/14622200410001669169. No abstract available. PMID 15203821
- [Derived] Berlin I, Singleton EG, Heishman SJ. Cross validation of the prognostic and diagnostic utility of tobacco craving in a general and a pregnant sample of treatment-seeking smokers. Drug Alcohol Depend. 2015 Sep 1;154:174-83. doi: 10.1016/j.drugalcdep.2015.06.034. Epub 2015 Jun 29. PMID 26160457
- [Derived] Berlin I, Grange G, Jacob N, Tanguy ML. Nicotine patches in pregnant smokers: randomised, placebo controlled, multicentre trial of efficacy. BMJ. 2014 Mar 11;348:g1622. doi: 10.1136/bmj.g1622. PMID 24627552